CLINICAL TRIAL: NCT05055466
Title: SARS-CoV-2 Infections in Children and Potential Fecal-oral Transmission
Brief Title: COVID-19: Infectious Potential of SARS-CoV-2 Intestinal Shedding in Pediatric Patients (INPOSIS)
Acronym: INPOSIS
Status: Completed | Type: Observational
Sponsor: St. Anna Kinderkrebsforschung (Other)
Responsible Party: Sponsor
Other Study IDs: INPOSIS
Record Dates: First submitted 2021-09-21; First posted 2021-09-24 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-04

CONDITIONS: SARS-CoV-2 Infection; Covid19; Intestinal Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Stool samples, swabs from the palms, nasopharyngeal swabs including swabs from the oral cavity and biomaterial stored in a biorepository, including stool specimens from paediatric patients who were hospitalized for a variety of indications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The clinical courses of COVID-19 in children are reportedly mild, and may therefore readily escape diagnosis. Prolonged intestinal virus shedding has been reported in children, thus rendering the pediatric population a potentially important source of virus transmission. However, the infectious potential of SARS-CoV-2 (severe acute respiratory syndrome coronavirus type 2) excreted in the stool has remained enigmatic.

The investigators hypothesize that stools carrying the virus can represent a source of infection, at least in a proportion of instances, and therefore intend to screen stools of children admitted to the hospital regardless of the indication in order to assess the frequency of intestinal virus excretion. The screening will be performed by validated RTQ-PCR (reverse transcription quantitative polymerase chain reaction) assays. In positive cases, stool extracts will be used to inoculate permissive cells (e.g. VeroE6) under BSL3 (Biosafety Level 3) conditions, and the infectious potential of the viruses will be determined. The readout will be based on the assessment of cell cytopathic effects and on the expression of subgenomic mRNA. it is expected to recruit ~100 patients for the study.

Additionally, the investigators will specifically examine children admitted to the hospital because of COVID-19, and will determine the temporal correlation between viral loads in the upper respiratory tract (URT) and serial stool specimens as well as swabs from the palms and from the oral cavity using RTQ-PCR. Longitudinal studies on the infectious potential of viruses from the URT and stool will be performed using the experimental approach outlined above. For this part of the study, is is intended to recruit ~100 children.

Furthermore, samples derived from >200 patients from our biorepository will be used.

The insights gained from the study will greatly expand the knowledge on the epidemiological and clinical significance of SARS-CoV-2 infections in children. If stools are identified as a potential source of infection, the data will have an important impact on safety measures in specific settings such as the kindergarten.

DETAILED DESCRIPTION:
Background:

Overt COVID-19 is reportedly far less frequent children. In a study from China, children <10 years of age represented only 0.9% and children between 10-19 years of age only 1.2% of the diagnostically confirmed cases1. Very similar data were published by the Italian registry, indicating 0.5% and 0.7%, respectively2. In the largest pediatric study published to date including >2000 children, 4% had asymptomatic courses, 90% had mild or moderate clinical courses, and severe manifestations were documented in 6% of cases, mostly involving infants below 1 year of age3. Some reports indicated asymptomatic courses in as many as 16-30% of affected children within individual age groups3,4. In addition to common symptoms such as fever and dry cough (40-100% of cases), diarrhea was a frequent observation in children with COVID-19 (10-30% of cases), in contrast to adults with overt disease (4% of cases) 5-11. Virus shedding into the stool was commonly observed in children for more than one month after resolution of acute infection7,10. However, the infectious potential of intestinal virus shedding, which has been demonstrated for the related viruses SARS-CoV and MERS-CoV (Middle East Respiratory syndrome coronavirus), is currently unclear for SARS-CoV-212,13. Due to the mild or even asymptomatic courses of COVID-19, children might represent an important source of disease transmission. With the increasing numbers of adults who are vaccinated and the appearance of new variants of the virus displaying different properties, the situation in children might certainly change and may need to be reevaluated. The proposed study in collaboration with different pediatric facilities in Austrian hospitals therefore offers an excellent opportunity to address different aspects of COVID-19 pertaining to the pediatric population.

Hypotheses:

* Shedding of SARS-CoV-2 into the stool is detectable in a proportion of asymptomatic children
* In patients with COVID-19, the frequency of intestinal virus excretion is higher and persists for prolonged time periods post infection
* Viruses excreted with the stool may display infectious potential

Study design:

During the study period of 12 months, it is intended to investigate ~500 pediatric patients admitted to the hospital for reasons unrelated to COVID-19, with the aim to screen for the occurrence of SARS-CoV-2 shedding into the stool in children who are not suspected to carry the virus. The indicated number of pediatric patients to be recruited is based on the maximum achievable number within the outlined study period. Currently, it is not possible to predict the proportion of patients with intestinal excretion of SARS-CoV-2. Additionally, the investigators will screen ~100 pediatric patients with COVID-19 to determine the frequency and duration of intestinal virus shedding. The majority of patients will only be investigated upon admission to the hospital and follow-up samples will be obtained in patients who tested positive at first analysis to document the duration of virus detectability. Furthermore, biomaterial stored in a biorepository, including stool specimens from pediatric patients who were hospitalized for a variety of indications, will be analyzed to determine the detectability of SARS-CoV-2 by molecular screening, and positive cases will be subjected to further analysis, as specified below.

Molecular testing of SARS-CoV-2 will be performed by a validated and certified RTQ-PCR assay established according to guidelines of the German reference center, the Robert Koch Institute in Berlin. Processing of clinical specimens will be carried out in line with pertinent biosafety regulations. The testing for infectious properties of SARS-CoV-2 pathogens detected in clinical specimens including particularly stool (and potentially nasopharyngeal swabs) will be carried out in a BSL3 facility (in collaboration with Prof. Dr. Willinger, Medical University of Vienna) by using permissive cell lines (VeroE6, CaCo2, or HCT116) under appropriate culture conditions. The readout will be based on the documentation of cell cytopathic effects and expression of subgenomic mRNA using established RTQ-PCR tests.

Sample collection and handling logistics:

Prospective analyses - stool samples (and various control specimens from other sites including swabs from the pharynx, oral cavity, nose, and palms) will be collected and stored at 4°C until transfer to the central laboratory, Labdia Labordiagnostik. The samples will be transferred in line with the biosafety regulations (UN3373) by a rapid delivery service (EMS or similar), to ensure arrival of the samples within three days (usually on the same day). Upon receipt, samples will be processed immediately (virus elution in phosphate buffered saline) and subjected to molecular analysis. In positive cases, stool extracts will be used as quickly as possible to inoculate permissive cells (e.g. VeroE6) under BSL3 safety conditions, and the infectious potential of the viruses will be determined. The readout will be based on the assessment of cell cytopathic effects and on the expression of subgenomic mRNA.Primary samples and isolated RNA will be stored at Labdia in a dedicated freezer at -80°C until the end of the study, and will be discarded thereafter.

Retrospective analyses - biomaterial that was collected and stored in a biorepository of Labdia Labordiagnostik

Ethical considerations and statistics:

Ethical approval for the study and informed consent for participation in the study from the patients and/or their legal representatives as well as the staff members has been obtained.

Personal data will be available exclusively in the certified clinical laboratory, Labdia Labordiagnostik, performing the diagnostic testing. Data processing for the present study will be done in a pseudonymized manner by assigning serial numbers.

In line with the principal aims of the study, Fisher´s exact test will be employed for comparing the incidence of SARS-CoV-2 detectability in pharyngeal and stool specimens, and for assessing the occurrence of infectious virus in stool specimens.

Expected outcome and future plans:

Due to the relative paucity of data on COVID-19 in specific pediatric settings, the proposed study will provide important insights into the clinically and epidemiologically relevant topics outlined above. The data obtained will serve as basis for ensuing large-scale studies addressing the infectious potential of intestinal shedding of the virus, and the measures required for various children facilities.

Testing for infectious properties of SARS-CoV-2 pathogens detected in clinical specimens including particularly stool (and potentially nasopharyngeal swabs) will be carried out by using permissive cell lines (VeroE6, CaCo2, or HCT116) under appropriate culture conditions. The readout will be based on the documentation of cell cytopathic effects and expression of subgenomic mRNA using established RTQ-PCR tests

In general, the collection of samples will be performed at a single time point in each patient, upon admission to the hospital. Within the prospective part of the study, follow-up samples will be collected from patients with COVID-19 displaying virus shedding into the stool. For the assessment of cytopathic effects and expression of subgenomic mRNA, fresh samples will be used, whenever possible. In all other instances, samples will be frozen at -80°C, and analyzed at a later point using an established protocol.

Clinical significance:

Due to the apparently common occurrence of prolonged intestinal SARS-CoV-2 shedding in children, who may not display any disease symptoms, it is of paramount importance to understand whether this putative way of virus transmission is of clinical and epidemiological relevance, as a basis for developing appropriate protection measures. Elucidation of the modes of transmission is critical for current and future approaches to the containment of SARS-CoV-2 spreading.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized pediatric patients: 0-18 years of age
* Informed consent for collection and retention of biomaterial

Exclusion Criteria:

* Absence of informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients admitted to the hospital for reasons unrelated to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Cytopathic effects and expression of subgenomic mRNA | A single time point in each patient, upon admission to the hospital
  Testing for infectious properties of SARS-CoV-2 pathogens detected in clinical specimens including particularly stool (and potentially swabs from the palms, nasopharyngeal swabs including swabs from the oral cavity) will be carried out by using permissive cell lines (VeroE6, CaCo2, or HCT116) under appropriate culture conditions. The readout will be based on the documentation of cell cytopathic effects and expression of subgenomic mRNA using established RTQ-PCR tests.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lion, Prof, MD, PhD, MSc, Study Chair — St.Anna Kinderkrebsforschung (CCRI); Meryl Haas, MSc, Principal Investigator — St.Anna Kinderkrebsforschung (CCRI)
Locations (4):
- Austria (4):
  - St.Anna Children´s Hospital, Vienna, Austria(AUT)
  - University Hospital Krems, Krems
  - University Hospital Tulln, Tulln
  - Klinik Ottakring, Vienna